CLINICAL TRIAL: NCT03323216
Title: BIO-2-HEART Study (Identifying New BIOmarkers in Patients With Type 2 Diabetes Mellitus and HEArt Failure Receiving Cardiac Resynchronization Therapy Device Implantation)
Brief Title: BIO-2-HEART: Identification of Biomarkers in T2DM and Heart Failure
Acronym: BIO-2-HEART
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Ben Kappel, Principal Investigator, RWTH Aachen University
Other Study IDs: 16-132
Record Dates: First submitted 2017-09-26; First posted 2017-10-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — Walk Test; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No diabetes: Patients without diabetes
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: Study specific questionnaire; Procedure: Blood collection
- Type 2 diabetes: Patients with diagnosis of type 2 diabetes (new/established)
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: Study specific questionnaire; Procedure: Blood collection
- Prediabetes: Patients with an intermediate state of hyperglycemia with glycemic parameters above normal but below the diabetes threshold.
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: Study specific questionnaire; Procedure: Blood collection

INTERVENTIONS:
Diagnostic Test: 6-minute walk test — The 6-minute walk test is a functional test established in the clinic to assess the performance of a patient. The patient walks continuously for 6 minutes without interruption as far as possible. Breaks, speed changes and running are allowed.
  Test is performed prior the intervention and 6 months after the intervention.
Diagnostic Test: Study specific questionnaire — Study specific questionnaire
  The questionnaire is performed prior and 6 months after the intervention.
Procedure: Blood collection — Blood collection during surgery:
  * coronary sinus
  * arterial
  * peripheral venous
  Blood collection 6 months after surgery:
  - peripheral venous

SUMMARY:
The primary aim of the current study is a better understanding of the role of Type 2 Diabetes Mellitus (T2DM) in heart failure and, in particular, changes in cardiac metabolism, which may contribute to heart failure. Various biomarkers in the coronary artery blood, as well as in the arterial and peripheral venous blood, are to be identified for this purpose. Included are patients with and without T2DM and with or without heart failure (HFpEF, HFmrEF, HFrEF), who have a clinically indicated and guidance-appropriate Cardiac Resynchronisation Therapy (CRT) implantation or pulmonary vein ablation/electrophysiological examination.

Not all patients currently benefit from the implantation of a CRT system (so-called non-responder). Despite narrow inclusion criteria, these "non-responders" cannot be unmasked in advance of the implantation. A further aim of this study is to identify biomarkers, which can be determined in advance of implantation to differentiate between responders and non-responders.

DETAILED DESCRIPTION:
The primary aim of the current study is a better understanding of the role of Type 2 Diabetes Mellitus (T2DM) in heart failure and, in particular, changes in cardiac metabolism, which may contribute to heart failure. Various biomarkers in the coronary artery blood, as well as in the arterial and peripheral venous blood, are to be identified for this purpose. Included are patients with and without T2DM, who have a clinically indicated and guidance-appropriate Cardiac Resynchronisation Therapy (CRT) implantation due to their cardiac insufficiency and patients who have a clinically indicated electrophysiological examination (EPU) or pulmonary vein ablation (PVI).

Not all patients currently benefit from the implantation of a CRT system (so-called non-responder). Despite narrow inclusion criteria, these "non-responders" cannot be unmasked in advance of the implantation. Thus, a further aim of this study is to identify biomarkers, which can be determined in advance of implantation to differentiate between responders and non-responders.

Patient selection is based on the previously defined inclusion and exclusion criteria. The patient is informed by the physician and gives written consent to participate in the study. Prior to the implantation of the CRT system/the electrophysiological examination(EPU)/pulmonary vein ablation(PVI), the patient first responds to a study-related questionnaire and performs a 6-minute walk test.

Afterwards the clinically indicated, elective CRT implantation/EPU/PVI is performed by experienced physicians of the Medical Clinic I. Routinely, an arterial pressure catheter for invasive blood pressure monitoring (usually arteria radialis) is inserted. In addition, 2 peripheral venous accesses are established. The system of the CRT system is carried out via a small pectoral section. The cardiac probes are inserted into the heart via the subclavian vein. First, the probe is implanted in the right ventricle and, if necessary, a probe is placed in the right atrium. For EPU/PVI a femoral vein acsess is established.

To establish the coronary sinus (CS) probe, the intubation of the coronary sinus is performed by means of a guide catheter, which can be used to take blood samples. After intubation of the coronary sinus, the coronary artery blood is taken from the guide catheter for the study as well as arterially via the underlying pressure catheter as well as peripheral venous over a horizontal venous catheter. During EPU/PVI the coronary sinus has also to be intubated due to the ablation protocol. The blood sampling does not take more than 1-2 minutes.

The surgery is then terminated as planned and postoperative care is performed according to the standard operation procedure (SOP) of the Medical Clinic I. Within the framework of a control visit routinely performed in the Medical Clinic I , an echocardiographic follow-up of heart failure, a history assessment and a laboratory-based blood analysis are performed 6 months after CRT implantation. In the context of this visit peripheral venous blood is collected again for the study. In addition, the 6-minute walk test is performed once more and the patient receives the same questionnaire again.

Laboratory routine blood analysis is performed in the central laboratory of the University Hospital of Aachen and is independent of the study. The analysis measures standard parameters such as electrolytes, blood count, retention parameters, glucose, HbA1c, liver values, N-terminal Brain Natriuretic Peptide (NT-pro-BNP) etc. .

A blood gas analysis of the study blood is performed out first. The remaining blood is processed and stored at -80 ° C, so-called "biobank", for further biomarker analysis, e.g. metabolite analysis, peptides/proteins and RNA.

ELIGIBILITY:
Inclusion Criteria:

1. guideline-appropriate clinical indication for CRT implantation/electrophysiologial examination/pulmonary vein ablation
2. age of majority
3. written declaration of consent
4. persons who are able to work and mentally able to follow the instructions of the study staff
5. free access routes

Exclusion Criteria:

1. anemia Hb <8 mg / dl
2. patients with acute infectious disease (e.g. pneumonia)
3. non-intubatable coronary sinus
4. patients who do not have access to the subclavian vein (e.g. thrombosis of the subclavian vein or superior vena cava)
5. patients with idiopathic hypertrophic, restrictive or constrictive cardiomyopathy, or heart failure due to a known inflammatory or infiltrating disease (e.g. amyloidosis, sarcoidosis) or a constrictive disease
6. patients with heart failure by sepsis
7. persons with acute myocardial ischaemia, e.g. by angina pectoris or ECG changes under load
8. patients with acute coronary syndrome are not implanted in the past 3 months
9. patients who were hospitalized during the last month due to heart failure and who had to be treated intravenously with diuretics or inotropic substances
10. patients with mechanical aortic valve or tricuspid valve
11. patients with heart transplant.
12. patients with acute liver or renal failure
13. pregnant and lactating women
14. patients placed under an official or judicial order in an institution
15. patients who are in a dependency or employment relationship with the sponsor or auditor
16. taking an investigational medicinal product 30 days before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without heart failure (HFrEF, HFmrEF, HFpEF) plus known status of type 2 diabetes (yes/no)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen partial pressure (pO2) [mmHg] | Directly prior to the CRT-implantation
  Results of blood gas analysis:
  Oxygen partial pressure (pO2) [mmHg]
Oxygen partial pressure (pO2) [mmHg] | 6 months after CRT-implantation
  Results of blood gas analysis:
  Oxygen partial pressure (pO2) [mmHg]
Carbon dioxide partial pressure (pCO2) [mmHg] | Directly prior to the CRT-implantation
  Results of blood gas analysis:
  Carbon dioxide partial pressure (pCO2) [mmHg]
Carbon dioxide partial pressure (pCO2) [mmHg] | 6 months after CRT-implantation
  Results of blood gas analysis:
  Carbon dioxide partial pressure (pCO2) [mmHg]
potential of hydrogen (pH) value [-] | Directly prior to the CRT-implantation
  Results of blood gas analysis:
  pH value [-]
potential of hydrogen (pH) value [-] | 6 months after CRT-implantation
  Results of blood gas analysis:
  pH value [-]
Base excess [mmol] | Directly prior to the CRT-implantation
  Results of blood gas analysis:
  Base excess [mmol]
Base excess [mmol] | 6 months after CRT-implantation
  Results of blood gas analysis:
  Base excess [mmol]
Lactate [mmol/l] | Directly prior to the CRT-implantation
  Results of blood gas analysis:
  Lactate [mmol/l]
Lactate [mmol/l] | 6 months after CRT-implantation
  Results of blood gas analysis:
  Lactate [mmol/l]
Glucose [mg/dl] | Directly prior to the CRT-implantation
  Results of blood gas analysis:
  Glucose [mg/dl]
Glucose [mg/dl] | 6 months after CRT-implantation
  Results of blood gas analysis:
  Glucose [mg/dl]
Electrolytes (K+, Na2+, Ca2+) [mmol/l] | Directly prior to the CRT-implantation
  Results of blood gas analysis:
  Electrolytes (K+, Na2+, Ca2+) [mmol/l]
Electrolytes (K+, Na2+, Ca2+) [mmol/l] | 6 months after CRT-implantation
  Results of blood gas analysis:
  Electrolytes (K+, Na2+, Ca2+) [mmol/l]
High-sensitive troponin T [µg/L] | Directly prior to the CRT-implantation
  Markers of myocardial ischemia and heart failure:
  High-sensitive troponin T [µg/L]
High-sensitive troponin T [µg/L] | 6 months after CRT-implantation
  Markers of myocardial ischemia and heart failure:
  High-sensitive troponin T [µg/L]
Total creatine kinase [µg/L] | Directly prior to the CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Total creatine kinase [µg/L]
Total creatine kinase [µg/L] | 6 months after CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Total creatine kinase [µg/L]
Creatinine kinase-myocardial band (CK-MB) [µg/L] | Directly prior to the CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Creatinine kinase-myocardial band (CK-MB) [µg/L]
Creatinine kinase-myocardial band (CK-MB) [µg/L] | 6 months after CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Creatinine kinase-myocardial band (CK-MB) [µg/L]
Aspartate aminotransferase [µg/L] | Directly prior to the CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Aspartate aminotransferase [µg/L]
Aspartate aminotransferase [µg/L] | 6 months after CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Aspartate aminotransferase [µg/L]
Lactate dehydrogenase [µg/L] | Directly prior to the CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Lactate dehydrogenase [µg/L]
Lactate dehydrogenase [µg/L] | 6 months after CRT-implantation
  Markers of myocardial ischemia and heart failure:
  Lactate dehydrogenase [µg/L]
N-terminal pro-B-type natriuretic peptide (NT-proBNP) [µg/L] | Directly prior to the CRT-implantation
  Markers of myocardial ischemia and heart failure:
  N-terminal pro-B-type natriuretic peptide (NT-proBNP) [µg/L]
N-terminal pro-B-type natriuretic peptide (NT-proBNP) [µg/L] | 6 months after CRT-implantation
  Markers of myocardial ischemia and heart failure:
  N-terminal pro-B-type natriuretic peptide (NT-proBNP) [µg/L]
High-sensitive C-reactive protein (CRP) [µg/L] | Directly prior to the CRT-implantation
  Cytokines and inflammation markers:
  High-sensitive C-reactive protein (CRP) [µg/L]
High-sensitive C-reactive protein (CRP) [µg/L] | 6 months after CRT-implantation
  Cytokines and inflammation markers:
  High-sensitive C-reactive protein (CRP) [µg/L]
Procalcitonin (PCT) [µg/L] | Directly prior to the CRT-implantation
  Cytokines and inflammation markers:
  Procalcitonin (PCT) [µg/L]
Procalcitonin (PCT) [µg/L] | 6 months after CRT-implantation
  Cytokines and inflammation markers:
  Procalcitonin (PCT) [µg/L]
Interleukin 6 (IL-6) [µg/L] | Directly prior to the CRT-implantation
  Cytokines and inflammation markers:
  Interleukin 6 (IL-6) [µg/L]
Interleukin 6 (IL-6) [µg/L] | 6 months after CRT-implantation
  Cytokines and inflammation markers:
  Interleukin 6 (IL-6) [µg/L]

CONTACTS AND LOCATIONS:
Overall Officials: Ben Kappel, MD PhD, Principal Investigator — Uniklinik RWTH Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Askoxylakis V, Thieke C, Pleger ST, Most P, Tanner J, Lindel K, Katus HA, Debus J, Bischof M. Long-term survival of cancer patients compared to heart failure and stroke: a systematic review. BMC Cancer. 2010 Mar 22;10:105. doi: 10.1186/1471-2407-10-105. PMID 20307299
- [Background] Bahtiyar G, Gutterman D, Lebovitz H. Heart Failure: a Major Cardiovascular Complication of Diabetes Mellitus. Curr Diab Rep. 2016 Nov;16(11):116. doi: 10.1007/s11892-016-0809-4. PMID 27730517
- [Background] Kappel BA, Marx N, Federici M. Oral hypoglycemic agents and the heart failure conundrum: Lessons from and for outcome trials. Nutr Metab Cardiovasc Dis. 2015 Aug;25(8):697-705. doi: 10.1016/j.numecd.2015.06.006. Epub 2015 Jun 18. PMID 26164634
- [Background] Sun H, Guan Y, Wang L, Zhao Y, Lv H, Bi X, Wang H, Zhang X, Liu L, Wei M, Song H, Su G. Influence of diabetes on cardiac resynchronization therapy in heart failure patients: a meta-analysis. BMC Cardiovasc Disord. 2015 Mar 21;15:25. doi: 10.1186/s12872-015-0018-0. PMID 25880202
- [Background] Watson CJ, Ledwidge MT, Phelan D, Collier P, Byrne JC, Dunn MJ, McDonald KM, Baugh JA. Proteomic analysis of coronary sinus serum reveals leucine-rich alpha2-glycoprotein as a novel biomarker of ventricular dysfunction and heart failure. Circ Heart Fail. 2011 Mar;4(2):188-97. doi: 10.1161/CIRCHEARTFAILURE.110.952200. Epub 2011 Jan 31. PMID 21282491
- [Background] Truong QA, Januzzi JL, Szymonifka J, Thai WE, Wai B, Lavender Z, Sharma U, Sandoval RM, Grunau ZS, Basnet S, Babatunde A, Ajijola OA, Min JK, Singh JP. Coronary sinus biomarker sampling compared to peripheral venous blood for predicting outcomes in patients with severe heart failure undergoing cardiac resynchronization therapy: the BIOCRT study. Heart Rhythm. 2014 Dec;11(12):2167-75. doi: 10.1016/j.hrthm.2014.07.007. Epub 2014 Jul 8. PMID 25014756
- [Background] Costello-Boerrigter LC, Lapp H, Boerrigter G, Lerman A, Bufe A, Macheret F, Heublein DM, Larue C, Burnett JC Jr. Secretion of prohormone of B-type natriuretic peptide, proBNP1-108, is increased in heart failure. JACC Heart Fail. 2013 Jun;1(3):207-12. doi: 10.1016/j.jchf.2013.03.001. Epub 2013 Jun 3. PMID 24621871
- [Background] Marques FZ, Vizi D, Khammy O, Mariani JA, Kaye DM. The transcardiac gradient of cardio-microRNAs in the failing heart. Eur J Heart Fail. 2016 Aug;18(8):1000-8. doi: 10.1002/ejhf.517. Epub 2016 Apr 12. PMID 27072074
- [Background] Bergman BC, Tsvetkova T, Lowes B, Wolfel EE. Myocardial glucose and lactate metabolism during rest and atrial pacing in humans. J Physiol. 2009 May 1;587(Pt 9):2087-99. doi: 10.1113/jphysiol.2008.168286. Epub 2009 Mar 16. PMID 19289551